CLINICAL TRIAL: NCT00449540
Title: Phase III Randomized Double-Blind Parallel Group Sham-Controlled Study Evaluating the Efficacy and Safety of Non-invasive Non-repetitive Transcranial Magnetic Stimulation (TMS) for the Acute Preemptive Treatment of the Aura Phase of Migraine Headache
Brief Title: Efficacy and Safety of TMS for the Preemptive Treatment of Migraine With Aura
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuralieve (Industry)
Responsible Party: Ting W. Lu / President and Chief Operating Officer, Neuralieve, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL-2006-001
Record Dates: First submitted 2007-03-18; First posted 2007-03-20 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-07

CONDITIONS: Migraine With Aura
Keywords: Migraine with aura; aura; TMS
MeSH Terms: conditions — Migraine with Aura; Epilepsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Transcranial Magnetic Stimulation (TMS) Device (Active Comparator): Both arms of participants receive identical looking devices and were instructed use the same treatment protocol. Participants in each group were instructed to treat with the device within one hour of onset of migraine aura.
  Interventions: Device: Active Transcranial Magnetic Stimulation (TMS) Device
- Sham TMS Device (Sham Comparator): Both arms of participants receive identical looking devices and were instructed use the same treatment protocol. Participants in each group were instructed to treat with the device within one hour of onset of migraine aura.
  Interventions: Device: Sham TMS Device

INTERVENTIONS:
Device: Active Transcranial Magnetic Stimulation (TMS) Device — Transcranial Magnetic Stimulation Device treatment
  Arms: Active Transcranial Magnetic Stimulation (TMS) Device
Device: Sham TMS Device — Simulated Sham treatment without TMS delivery
  Arms: Sham TMS Device

SUMMARY:
Assess safety and efficacy of Transcranial Magnetic Stimulation (TMS) for the treatment of migraine with aura

The hypothesis is that TMS treatments delivered to the occipital cortex of the brain can stop or interrupt the spreading cortical brain activity that causes or contributes to the migraine headache. Two TMS treatments at an intensity of <1 Tesla for ~500 microseconds, approximately 30 seconds apart, may stop the aura and prevent the subsequent headache.

DETAILED DESCRIPTION:
In the Lead-in Phase participants will use a Personal Digital Assistant (PDA) to keep an electronic diary of their migraine episodes. During a migraine episode, as well as the time in between headaches, the PDA prompts the participant to answer questions. Each evening, the participant will place the PDA into an electronic telephone cradle, and the information will be transmitted electronically from the PDA to the data management team to assess the frequency of migraine episodes and participant proficiency with the PDA. During this one month period, the participant must experience at least one migraine with aura episode to enter the Treatment Phase.

After one month, the participant will return to the clinic with their PDA and will enter the Treatment Phase to be randomized to either the TMS only group or the Sham stimulation only group. Participant will enter information into the PDA for three migraine auras treated or three months, which ever comes first.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years
* Will comply with requirements of the protocol
* Have a consistent history of migraine with visual aura of at least one year

  •>30% of episodes have a visual aura preceding headaches
* Approximately 90% of the time have moderate or severe headaches following their aura
* Fulfills the International Classification of Headache Disorders, 2nd Edition(ICHD-II) criteria(for migraine headache with aura after administration of a clinical interview by study personnel
* Has a history of 1-8 migraine headache episodes with aura per month
* Can differentiate a migraine headache from other types of headaches
* Participant is post-menopausal, sterilized, not breastfeeding, her pregnancy test is negative

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Routinely experiences any other type of headache that would confound discrimination from migraine headache with aura
* Have migraine with prolonged aura > 60 minutes
* Have headaches due to other underlying pathology
* Have headaches related to head or neck trauma
* Overuse headache medications:
* Has an intracranial metallic or Transcranial Magnetic Stimulation (TMS) implant or other metallic implants
* Has cardiac pacemaker or any other implanted electronic device
* Has any known history of alcohol abuse, drug dependency, or significant psychiatric illness in the previous 12 months
* Having any medical condition, including but not limited to: clinically significant renal or hepatic disease; uncontrolled hypertension; clinically significant coronary vascular disease not stable for the past 6 months; personal or family history of seizures or taking medications for seizures or drugs that may lower seizure threshold, cerebral vascular ischemia; infarct; hemorrhage, or other central nervous system disease (e.g., multiple sclerosis, amyotrophic lateral sclerosis); unstable metabolic disease, hypoglycemia or diabetes; malignancy within the past 5 years excluding cutaneous basal cell carcinoma; tuberculosis
* Has participated in any other investigational study within the previous 30 days.
* Cannot place the device within 1 cm of the scalp.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Lipton, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (14):
- United States (14):
  - San Francisco Headache Clinic, San Francisco, California
  - Mile High Research Center, Denver, Colorado
  - Diamond Headache Clinic, LTD, Chicago, Illinois
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Westside Family Medical Center, Kalamazoo, Michigan
  - Clinvest, Inc., Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Kirchner Headache Clinic, Omaha, Nebraska
  - Montefiore Headache Center, The Bronx, New York
  - The Ohio State University, Columbus, Ohio
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Nashville Neuroscience Group, Nashville, Tennessee
  - The Innovative Clinical Research Center, Alexandria, Virginia
  - Swedish Headache Center, Seattle, Washington

REFERENCES:
- [Derived] Lipton RB, Dodick DW, Silberstein SD, Saper JR, Aurora SK, Pearlman SH, Fischell RE, Ruppel PL, Goadsby PJ. Single-pulse transcranial magnetic stimulation for acute treatment of migraine with aura: a randomised, double-blind, parallel-group, sham-controlled trial. Lancet Neurol. 2010 Apr;9(4):373-80. doi: 10.1016/S1474-4422(10)70054-5. Epub 2010 Mar 4. PMID 20206581

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 267 participants enrolled in the 30 day Lead-In phase as described. 66 participants did not experience migraine in the 30 days allotted and therefore were not moved to the treatment phase. 201 participants were moved to the treatment phase
Groups:
- 30 Day Lead in Phase: some particpants did not experience migrain in the 30 days allotted and therefore were not moved to the treatment phase
- Active TMS: Active Transcranial Magnetic Stimulation Device
- Sham TMS Device: Device which does not deliver TMS pulse
Period: Pretreatment Phase
Arm/Group | 30 Day Lead in Phase | Active TMS | Sham TMS Device
Started | 267 | 0 | 0
Completed | 201 | 0 | 0
Not Completed | 66 | 0 | 0
Not completed — No migraine experienced | 66 | 0 | 0
Period: Treatment Phase
Arm/Group | 30 Day Lead in Phase | Active TMS | Sham TMS Device
Started | 0 | 102 | 99
Completed | 0 | 82 | 82
Not Completed | 0 | 20 | 17
Not completed — did not experience or treat migraine | 0 | 20 | 17

BASELINE CHARACTERISTICS:
Groups:
- Active Transcranial Magnetic Stimulation (TMS) Device: Active Transcranial Magnetic Stimulation Device Treatment
- Sham TMS Device: Simulated Sham treatment without TMS
- Total: Total of all reporting groups
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Device | Sham TMS Device | Total
Number analyzed (Participants) | 102 | 99 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 102 | 99 | 201
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (11.2) | 40.1 (10.83) | 39.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 78 | 158
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 102 | 99 | 201

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing no Pain at Two Hours Post-treatment
Description: Number of participants experiencing no pain at two hours post-treatment divided by total number of participants treated. For each treated aura episode during the migraine treatment phase, the subjects rated the pain intensity of their headache as none, mild, moderate or severe at baseline (before application of the study device) at 30 minutes, and at 1, 2, 24, and 48 hours posttreatement.
Time Frame: Two hours
Population: Full-analysis set: intention to treat population (201) adjusted for those participants who did not administer treatment during the study period
Measure: Number; unit: percentage of participants
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Device | Sham TMS Device
Number analyzed (Participants) | 82 | 82
percentage of participants | 39 | 22

2. Secondary Outcome: Percentage of Participants Who Have Symptoms of Nausea
Description: Percentage of participants who have symptoms of nausea two hours post treatment. For each treated aura episode, the subjects rated the severity of photophobia, nausea, and phonophobia as none, mild, moderate, or severe at baseline and recorded the presence or absence of vomiting at baseline (before application of the device) at 30 minutes, and at 1, 2, 24 and 48 hours posttreatment.
Time Frame: two hours post treatment
Measure: Number; unit: percentage of participants
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Device | Sham TMS Device
Number analyzed (Participants) | 82 | 82
percentage of participants | 38 | 40

3. Secondary Outcome: Percentage of Participants Who Have Symptoms Phonophobia
Description: Percentage of participants who have symptoms of phonophobia two hours post treatment. For each treated aura episode, the subjects rated the severity of photophobia, nausea, and phonophobia as none, mild, moderate, or severe at baseline and recorded the presence or absence of vomiting at baseline (before application of the device) at 30 minutes, and at 1, 2, 24 and 48 hours posttreatment.
Time Frame: 2 hours post treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Device | Sham TMS Device
Number analyzed (Participants) | 82 | 82
Percentage of Participants | 57 | 63

4. Secondary Outcome: Percentage of Participants Who Have Photophobia
Description: Percentage of participants who have symptoms of photophobia two hours post treatment. For each treated aura episode, the subjects rated the severity of photophobia, nausea, and phonophobia as none, mild, moderate, or severe at baseline and recorded the presence or absence of vomiting at baseline (before application of the device) at 30 minutes, and at 1, 2, 24 and 48 hours posttreatment.
Time Frame: 2 hours post treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Device | Sham TMS Device
Number analyzed (Participants) | 82 | 82
Percentage of participants | 70 | 78

ADVERSE EVENTS:
Groups:
- Active TMS Device - Treatment Related: Active Transcranial Magnetic Stimulation Device Treatment - Treatment related
- Sham TMS Device - Treatment Related: Simulated Sham treatment without TMS
- Active TMS - Not Treatment Related: Active Transcranial Magnetic Stimulation Device Treatment - Not treatment related
- Sham TMS Device - Not Treatment Related: Sham TMS Device - events that are not treatment related
Arm/Group | Active TMS Device - Treatment Related | Sham TMS Device - Treatment Related | Active TMS - Not Treatment Related | Sham TMS Device - Not Treatment Related
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/99 | 1/102 | 0/99
Other Adverse Events (participants affected / at risk) | 7/102 | 2/99 | 12/102 | 8/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS Device - Treatment Related (N=102) | Sham TMS Device - Treatment Related (N=99) | Active TMS - Not Treatment Related (N=102) | Sham TMS Device - Not Treatment Related (N=99)
optic neuritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One serious adverse event,optic neuritis,was reported in one subject who was randomized to the TMS group. The optic neuritis for Subject was not considered by the investigator and medical monitor to be related to the study treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS Device - Treatment Related (N=102) | Sham TMS Device - Treatment Related (N=99) | Active TMS - Not Treatment Related (N=102) | Sham TMS Device - Not Treatment Related (N=99)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizzines (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tempromandibular joint syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Road traffic Accident (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less